CLINICAL TRIAL: NCT01565876
Title: Auxiliary Device to Alleviate Soldiers' Backload
Acronym: minkal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: Principal Investigator, amit druyan, The Institute of Military Physiology, Medical Corps, Israel Defense Force
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 963-2010-CLIL
Record Dates: First submitted 2011-07-04; First posted 2012-03-29 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Physiological Strain of Weight Bearing.
Keywords: weight bearing; physiological load

ARMS (1):
- study (Experimental): The participants will undergo 6 days of study. The first day of the study include medical examination, maximal oxigen consumption day and anthropometric mesurments.
  Then The participants will undergo heat tolerance test 5 times (in different days).
  first day- without load. second day- with back load of 40% of the body weight. third day- with back load of 40% of the body weight and the Auxilairy Device. fourth day- with back load of 60% of the body weight. fifth day- with back load of 60% of the body weight and the Auxilairy Device. The rectal temperature, skin teperature and heart rate will be mesured each day and compered afterwards.
  Interventions: Device: "Minkal"- Auxiliary device to alleviate backload

INTERVENTIONS:
Device: "Minkal"- Auxiliary device to alleviate backload — The participants will undergo 6 days of study. The first day of the study include medical examination, maximal oxigen consumption day and anthropometric mesurments.
  Then The participants will undergo heat tolerance test 5 times (in different days).
  first day- without load. second day- with back load of 40% of the body weight. third day- with back load of 40% of the body weight and the Auxilairy Device. fourth day- with back load of 60% of the body weight. fifth day- with back load of 60% of the body weight and the Auxilairy Device. The rectal temperature, skin teperature and heart rate will be mesured each day and compered afterwards.

SUMMARY:
Combat soldiers are required to perform under strenuous physical conditions; hence, their physical fitness is a crucial factor in their survivability.

The Auxiliary Device- "Minkal", is suggested (by its manufactures) to be able to reduce the soldiers' physiological strain by lowering the absolute load being carried by the soldier. As a result, it may improve the soldier's physiological abilities and performance through enduring missions with heavy loads, and may lead to better protection on the soldier from overuse injuries.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without any of the following: chronic background diseases, cardiovascular, lung or respiratory, heat stroke history, headaches,psychiatric background, musculoskeletal problems, and without drugs use.
* Lack of any acute disease during 2 weeks prior the study.
* Subjects will give their written consent for participating the study after being informed by the study's physician about the study's aims, importance and the possible risks.

Exclusion Criteria:

* Rectal temperature above 39 Celsius degrees.
* HR above maximal HR ( calculated as 220-age)
* The subject's will to stop the test.
* The researcher's/doctor's judgment.

Ages: 21 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Physiological Load with and without the auxiliary device | 6 days for each patient.
  The physiological load will be measured using a heat tolerance test(HTT). Each paricipant will undergo a HTT 5 times (in different days). first day- without load. second day- with back load of 40% of the body weight. third day- with back load of 40% of the body weight and the Auxilairy Device. fourth day- with back load of 60% of the body weight. fifth day- with back load of 60% of the body weight and the Auxilairy Device. The rectal temperature, skin teperature and heart rate will be mesured in each HTT and compered afterwards to assess the physiological load.

SECONDARY OUTCOMES:
Rectal temperature | 6 days
  The Rectal temperature will be mesured by a rectal thermistore during each HTT.
Skin temperature | 6 days
  The Skin temperature will be mesured by skin thermistores on three sites (chest, leg and arm).
Heart Rate | 6 days
  Heart rate will be monitored using a polar watch.
Sweat Rate | 6 days
  Sweat rate will be calculated from the patient's weight and his water balance.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Makernatz, MD, Principal Investigator — Institute physician; Yuval Heled, PhD, Study Director — Director of the military physiology institute, IDF medical corps; Ran Yanovich, MA, Study Director — The director's deputy of the military physiology institute, IDF medical corps
Locations (1):
- Institute of military physiology, Ramat Gan, Israel